CLINICAL TRIAL: NCT02008383
Title: Cabozantinib (XL184) With Panitumumab in Subjects With KRAS Wild-Type Metastatic Colorectal Cancer and Cabozantinib Monotherapy in Subjects With MET Amplified Treatment-Refractory Colorectal Cancer
Brief Title: Cabozantinib and Panitumumab to Treat KRAS Wild-Type Metastatic Colorectal Cancer
Acronym: CaboMAb
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Strickler, M.D. (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, John Strickler, M.D., Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00049983
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Panitumumab; Cabozantinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib and Panitumumab (Experimental): 60 mg Cabozantinib PO daily and 6 mg/kg Panitumumab IV every 2 weeks.
  Interventions: Biological: Panitumumab; Drug: Cabozantinib
- Cabozantinib (Experimental): 60 mg Cabozantinib PO daily.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Biological: Panitumumab — The FDA approved dose for panitumumab is 6mg/kg IV, every two weeks. This is the dose and schedule that will be used in this study.
  Other Names: Vectibix
  Arms: Cabozantinib and Panitumumab
Drug: Cabozantinib — There will be three parts to this phase I study: 1) the Combination Dose Finding cohort; 2) the Combination Expansion cohort; and 3) the Monotherapy MET Amplified cohort.
  Cabozantinib will start at a dose of 60 mg daily with reductions to 40 and 20 mg daily possible in the dose finding cohort. The combination expansion cohort dose will determined by the dose finding cohort. The Monotherapy MET Amplified cohort will recieve 60 mg Cabozantinib daily.
  Other Names: Cometriq

SUMMARY:
There will be three parts to this phase I study: 1) the Combination Dose Finding cohort; 2) the Combination Expansion cohort; and 3) the Monotherapy MET Amplified cohort. In the Combination Dose Finding cohort and the Combination Expansion cohort, we will combine cabozantinib and panitumumab in patients with KRAS wild-type metastatic colorectal cancer (CRC). In the Monotherapy MET Amplified cohort, we will screen at least 50 patients for MET gene amplification ("MET amplification"). Patients with MET amplification will receive cabozantinib only (monotherapy).

The primary objective of this open-label phase Ib trial are:

1. To determine the maximum tolerated dose and the recommended phase II dose for the combination of cabozantinib and panitumumab in patients with KRAS wild-type metastatic colorectal cancer and
2. To identify the objective response rate (ORR) of cabozantinib monotherapy in patients with prospectively identified MET amplified metastatic colorectal cancer.

The secondary objectives are:

1. To describe the non-dose limiting toxicities of cabozantinib and panitumumab.
2. To describe the clinical activity (ORR, PFS, OS) of cabozantinib and panitumumab.
3. To describe the safety and tolerability of cabozantinib monotherapy in patients with MET amplified colorectal cancer.
4. To describe the clinical activity (PFS, OS) of cabozantinib monotherapy in patients with MET amplified colorectal cancer.

ELIGIBILITY:
MET Amplification Screening Test Inclusion Criteria:

1. Histologically and/or cytologically confirmed and radiographically measurable KRAS wild-type adenocarcinoma of the colon or rectum that is metastatic and/ or unresectable. Subjects must have been treated with a fluoropyrimidine (e.g., 5-fluorouracil or capecitabine), oxaliplatin, irinotecan and bevacizumab or have contraindication to such treatment.
2. Prior treatment with anti-EGFR therapy (either panitumumab or cetuximab).
3. At least one site of disease that is measurable by RECIST (version 1.1) criteria that has not been previously irradiated; if the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Life expectancy greater than 3 months.
7. Capable of understanding and complying with the protocol requirements and has signed the informed consent document.
8. Adequate organ and marrow function as defined below:

Absolute neutrophil count ≥ 1,000/μl without colony stimulating factor support

Platelets ≥ 75,000/μl

Hemoglobin ≥ 8 g/dL

AST/ALT ≤ 3 X upper limit of normal (ULN)

Total bilirubin ≤ 1.5 X upper limit of normal (ULN)

Serum albumin ≥ 2.5 g/dL

MET Amplification Screening Test Exclusion Criteria:

1. Presence of or known history of brain/ CNS tumor or metastases.
2. KRAS exon 2 (codons 12 or 13) mutation detected in tumor tissue specimen.
3. Concurrent severe and/or uncontrolled medical conditions which may compromise participation in the study, including impaired heart function or clinically significant heart disease.
4. Concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic LMWH are permitted.
5. Previously experienced any of the following:

   1. clinically significant gastrointestinal bleeding within the last 6 months
   2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within the last 3 months
   3. any other signs indicative of pulmonary hemorrhage within the last 3 months
6. Radiographic evidence of cavitating pulmonary lesion(s).
7. Tumor in contact with, invading or encasing any major blood vessels.
8. Evidence of endotracheal or endobronchial tumor.
9. Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   1. Cardiovascular disorders including:

   i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening

ii. Any history of congenital long QT syndrome

iii. Any of the following within the last 6 months:

1. unstable angina pectoris
2. clinically-significant cardiac arrhythmias
3. stroke (including TIA, or other ischemic event)
4. myocardial infarction
5. thromboembolic event requiring therapeutic anticoagulation Note: Subjects with a venous filter (e.g., vena cava filter) are not eligible for this study.

   b. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including: i. Any of the following within the last 28 days:

<!-- -->

1. active peptic ulcer disease
2. active inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
3. malabsorption syndrome

ii. Any of the following within the last 6 months:

1. abdominal fistula
2. gastrointestinal perforation
3. bowel obstruction or gastric outlet obstruction
4. intra-abdominal abscess

Note: Complete resolution of an intra-abdominal abscess must be confirmed prior even if the abscess occurred more that 6 months ago.

c. Other disorders associated with a high risk of fistula formation or wound healing complications, including percutaneous endoscopic gastrostomy (PEG) tube placement within the last 3 months.

d. History of chronic pancreatitis.

10. Unable to swallow tablets.

11. Evidence within the last 2 years of another malignancy which required systemic treatment.

12. Known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.

Main Study Inclusion Criteria:

1. For the Monotherapy MET Amplified cohort only: MET gene amplification by prospective screening assay from peripheral blood.
2. Histologically and/or cytologically confirmed and radiographically measurable KRAS wild-type adenocarcinoma of the colon or rectum that is metastatic and/ or unresectable. Subjects must have been treated with a fluoropyrimidine (e.g., 5-fluorouracil or capecitabine), oxaliplatin, irinotecan and bevacizumab or have contraindication to such treatment. In addition, for the monotherapy MET Amplified cohort, must have received prior treatment with anti-EGFR therapy (either panitumumab or cetuximab).
3. At least one site of disease that is measurable by RECIST (version 1.1) criteria that has not been previously irradiated; if the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy greater than 3 months.
7. Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).
8. Women of childbearing potential must have a negative pregnancy test within 7 days before the first dose of study treatment.
9. Capable of understanding and complying with the protocol requirements and has signed the informed consent document.
10. Adequate organ and marrow function as defined by protocol.

Main Study Exclusion Criteria:

1. Cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/ mitomycin C within 6 weeks before the first dose of study treatment.
2. Prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment.
3. For Combination Dose Finding and Combination Expansion cohorts only: History of hypersensitivity reactions/anaphylaxis attributed to humanized and/or chimeric monoclonal antibodies or other such proteins. Hypersensitivity reactions that are clearly related to cetuximab may be permitted at the discretion of the Lead PI.
4. Radionuclide treatment, including yttrium-90 treatment, within 6 weeks of the first dose of study treatment.
5. Radiation therapy:

   a. to the thoracic cavity, abdomen or pelvis within 3 months of the first dose of study treatment or has ongoing complications or is without complete recovery and healing from prior radiation therapy b. to bone metastases within 14 days of the first dose of study treatment c. to any other site(s) within 28 days of the first dose of study treatment
6. Any other type of investigational agent within 28 days before the first dose of study treatment.
7. Not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia, oxaliplatin-related neuropathy, and other non-clinically significant adverse events.
8. Presence of or known history of brain/ CNS tumor or metastases.
9. KRAS exon 2 (codons 12 or 13) mutation detected in tumor tissue specimen.
10. Concurrent severe and/or uncontrolled medical conditions which may compromise participation in the study, including impaired heart function or clinically significant heart disease.
11. Prothrombin time (PT) or partial thromboplastin time (PTT) test ≥ 1.3 x laboratory upper limit of normal (ULN) within 7 days before the first dose of study treatment.
12. Concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic LMWH are permitted.
13. Chronic concomitant treatment of strong CYP3A4 inducers or CYP3A4 inhibitors.
14. Previously experienced any of the following:

    1. clinically significant gastrointestinal bleeding within 6 months before the first dose of study treatment
    2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment
    3. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
15. Radiographic evidence of cavitating pulmonary lesion(s).
16. Tumor in contact with, invading or encasing any major blood vessels.
17. Evidence of endotracheal or endobronchial tumor.
18. Uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    1. Cardiovascular disorders including:

    i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening

ii. Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment

iii. Any history of congenital long QT syndrome

iv. Any of the following within 6 months before the first dose of study treatment:

1. unstable angina pectoris
2. clinically-significant cardiac arrhythmias
3. stroke (including TIA, or other ischemic event)
4. myocardial infarction
5. thromboembolic event requiring therapeutic anticoagulation

   Note: Subjects with a venous filter (e.g., vena cava filter) are not eligible for this study.

   b. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

   i. Any of the following within 28 days before the first dose of study treatment

<!-- -->

1. active peptic ulcer disease
2. active inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
3. malabsorption syndrome

ii. Any of the following within 6 months before the first dose of study treatment:

1. abdominal fistula
2. gastrointestinal perforation
3. bowel obstruction or gastric outlet obstruction
4. intra-abdominal abscess

Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months before the first dose of study treatment.

c. Other disorders associated with a high risk of fistula formation or wound healing complications, including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy.

d. History of chronic pancreatitis.

e. Other clinically significant disorders such as:

i. active infection requiring IV antibiotic within 28 days before the first dose of study treatment

ii. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment

iii. history of organ transplant

iv. concurrent uncompensated hypothyroidism or thyroid dysfunction

Note: Patients with newly diagnosed thyroid conditions may participate if stable on a new regimen for at least 7 days before the first dose of study treatment.

v. history of surgery as follows:

1. major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
2. minor surgery, including dental procedures, within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications

In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery.

19. History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan.

20. Unable to swallow tablets.

21. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before start of treatment. Note: At baseline (i.e. screening), three ECGs to be obtained within 30 minutes but approximately 2 minutes apart (i.e. triplicate). If the average of the three consecutive results for QTcF is ≤ 500 ms, the subject meets eligibility in this regard.

22. Pregnant or breastfeeding.

23. For the Combination Dose Finding and Combination Expansion cohorts only: Previously identified allergy or hypersensitivity to components of the study treatment formulation or panitumumab.

24. Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

25. Evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment.

26. Known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2018-05-10 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RPTD) for the combination of cabozantinib and panitumumab | RPTD for the study will be determined at the completion of Phase I dose escalation cohort; estimated as 1 year
Objective response rate (ORR) of cabozantinib monotherapy in patients with prospectively identified MET amplified metastatic colorectal cancer | Approximately every 8 weeks and/or restaging

SECONDARY OUTCOMES:
Non-dose limiting toxicities of cabozantinib and panitumumab. | Continuous, every 4 weeks minimum until end of study estimated at 4 years
  Adverse events will be recorded
Response rate of cabozantinib and panitumumab | approximately every 8 weeks and/or restaging
  Response is assessed at restaging, approximately every 8 weeks.
Progression free survival associated with the cabozantinib and panitumumab regimen | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival associated with the cabozantinib and panitumumab regimen | From date of randomization until the date of death from any cause assessed up to 60 months
Progression free survival associated with cabozantinib monotherapy in patients with MET amplified colorectal cancer | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival associated with cabozantinib monotherapy in patients with MET amplified colorectal cancer | From date of randomization until the date of death from any cause assessed up to 60 months
To describe the safety and tolerability of cabozantinib monotherapy in patients with MET amplified colorectal cancer | Continuous, every 4 weeks minimum until end of study estimated at 4 years
  Adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: John Strickler, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Strickler JH, Rushing CN, Uronis HE, Morse MA, Niedzwiecki D, Blobe GC, Moyer AN, Bolch E, Webb R, Haley S, Hatch AJ, Altomare IP, Sherrill GB, Chang DZ, Wells JL, Hsu SD, Jia J, Zafar SY, Nixon AB, Hurwitz HI. Cabozantinib and Panitumumab for RAS Wild-Type Metastatic Colorectal Cancer. Oncologist. 2021 Jun;26(6):465-e917. doi: 10.1002/onco.13678. Epub 2021 Feb 9. PMID 33469991
- [Derived] Jia J, Howard L, Liu Y, Starr MD, Brady JC, Niedzwiecki D, Strickler JH, Nixon AB. Cabozantinib with or without Panitumumab for RAS wild-type metastatic colorectal cancer: impact of MET amplification on clinical outcomes and circulating biomarkers. Cancer Chemother Pharmacol. 2022 Mar;89(3):413-422. doi: 10.1007/s00280-022-04404-8. Epub 2022 Feb 16. PMID 35171350